CLINICAL TRIAL: NCT02291497
Title: Non-interventional, Prospective, Single-center Investigation With Exploratory Data Analysis to Delineate the Variability and Frequency of Symptoms and Disease Manifestations in Adult HPP Patients
Brief Title: Burden of Disease in Hypophosphatasia (HPP)
Status: Completed | Type: Observational
Sponsor: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Lothar Seefried, Dr. med., Wuerzburg University Hospital
Other Study IDs: HPP-Study
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Hypophosphatasia
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be stored till 2031
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypophosphatasia (HPP) is a rare, inherited metabolic disease caused by inactivating mutations in the Alkaline Phosphatase (ALPL) gene, coding for the Tissue-nonspecific alkaline phosphatase (TNAP). Penetrance and disease severity is very heterogenous, ranging from stillbirth to adult-onset manifestations. Especially the latter are again characterized by an extremely broad spectrum of symptoms. This scope of variability makes it difficult to attribute individual patients' symptoms to the disease and distinguish them from HPP independent health issues. Especially in adult HPP patients, musculoskeletal problems, including (fragility-) fractures / bone bruise, joint pain, reduced mobility, muscular weakness and pain and reduced muscular endurance appear to reflect the prevailing burden of disease, especially with respect these patients dis-abilities of daily life.

To expand current knowledge of the natural history of the disease as well as on disease specific musculoskeletal deficits in HPP, all adult patients with established Diagnosis of HPP known at the Orthopedic Institute, University of Würzburg, will be offered to participate in a single, multimodal assessment of their disease history, current symptoms and disabilities, lab evaluations and clinical and technical analysis of their musculoskeletal status and capabilities.

Patients will be invited to a day long visit to the clinic in order to perform the following assessments:

A) Epidemiologic / anamnestic information B) Physical examination C) Structured questionnaires D) Laboratory examinations E) Clinical functional testing F) Technical Examinations

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females (age ≥ 18 years)
* Established diagnosis of Hypophosphatasia
* Reduced Serum/Plasma ALP (Alkaline phosphatase)-Activity below age and sex specific reference range of the respective test kit applied (measured at least twice with a minimum 4 week interval)
* At least one of the items below:

  * Genetically secured ALPL-Mutation
  * Elevated PLP (Pyridoxal 5-Phosphate) (urine or serum), above ULN (Upper level of normal)
  * Symptoms of the disease
* Signed informed consent

Exclusion Criteria:

* Current / previous treatment with Asfotase alfa
* Current participation in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: see "Eligibility Criteria"
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Frequencies of main disease symptoms and main disease manifestations | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Unit, Orthopaedische Klinik Koenig-Ludwig-Haus, Lehrstuhl der Universitaet Wuerzburg, Würzburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Weider M, Schlagenhauf U, Seefried L. Oral health status of adult hypophosphatasia patients: A cross-sectional study. J Clin Periodontol. 2022 Dec;49(12):1253-1261. doi: 10.1111/jcpe.13718. Epub 2022 Sep 7. PMID 36054522